CLINICAL TRIAL: NCT03478306
Title: Diabetic Retinopathy: Effects of Melatonin Treatment on Visual Functions and Circadian Rhythm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Shakoor Ba-Ali, Principal Investigator, Medical Doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DR2; 2015-003955-23 (EudraCT Number)
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Retinopathy; Melatonin; Circadian Dysrhythmia; Circadian Rhythm Sleep Disorder, Unspecified Type
MeSH Terms: conditions — Diabetic Retinopathy; Sleep Disorders, Circadian Rhythm | interventions — Melatonin; Tablets

STUDY DESIGN:
Intervention Model Description: A Double-blind, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Melatonin and placebo tablets are identicle in terms of taste, colour, tablet-size etc. The tablets are packed and masked by external manufacturer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Melatonin, 1 tablet (4 mg), every evening 2 hours before bed in 21 days.
  Interventions: Drug: Melatonin 4 mg Tablet
- Arm 2 (Placebo Comparator): Place, 1 tablet (4 mg), every evening 2 hours before bed in 21 days.
  Interventions: Drug: Melatonin 4 mg Tablet

INTERVENTIONS:
Drug: Melatonin 4 mg Tablet — Participants are randomized into arm 1 or arm2, recieving melatonin or placebo, respectively, for 21 days, followed by 1 week of washout, and then swichting to the contralateral treatment arm.

SUMMARY:
This study evaluates the effect of melatonin 4 mg on circadian rhythm and visual function of patients with diabetes mellitus. Half of the patients will receive melatonin (arm-1) and the other half will receive placebo (arm-2), both groups in 3 weeks. After a week of washout, the patients will cross over to the other treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients
* Age range 40-75 years
* Participant should be legally competent

Exclusion Criteria:

* Other known eye disease.
* Eye disease manifestation during ocular examination.
* Competing neurologic and systemic conditions affecting retina.
* Use of any drugs influencing pupillary light reflex and sleep pattern.
* Refractive error with need of > 6 diopter lenses.
* Pregnancy
* Alcohol consumption during the trial
* Lack of cooperation
* Allergy to melatonin and/or preservatives in melatonin and placebo
* Reduced hepatic function
* Fluvoxamin intake due to drug interaction
* Consumption of Alpha-1 and beta-1 adnergic antagoists.
* Alcohol consumption during treatment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
Progression of diabetic retinopathy, oscillary potential | 3 weeks
  Progression of diabetic retinopati measured with electroretinography

SECONDARY OUTCOMES:
Post-illumination pupillary light response | 3 weeks
  Melanopsin-mediated pupillary response
Circadian photoentrainment | 3 weeks
  Salivary melatonin level and sleep assessment
Retinal structure | 3 weeks
  Retinal structure assessed by optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Shakoor Ba-Ali, Principal Investigator — Department of Ophthalmology, Rigshospitalet-Glostrup
Locations (1):
- Department of Ophthalmology, Rigshospitalet-Glostrup, Glostrup Municipality, RegionH, Denmark

IPD SHARING:
Plan to Share IPD: No